CLINICAL TRIAL: NCT04188275
Title: CIRCULATING MICRO-RNA (miRNA) AND AR-V7 MUTATIONAL STATUS IN METASTATIC CASTRATION-RESISTANT PROSTATE CANCER (CRPC): PRIMERA+ STUDY (PROSTATE CANCER INNOVATING MARKERS OF EXPECTED RESPONSE TO AGONIST LHRH+ ANDROGEN RECEPTOR INHIBITION
Acronym: PRIMERA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: PRIMERA
Record Dates: First submitted 2019-12-04; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: D011471; D064129; D035683; D009360; D014408
Keywords: Prostate Cancer; Metastatic Castration-Resistant; Biomarker Tumor
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Metastatic Castration Resistant Prostate Cancer: Metastatic Castration Resistant Prostate Cancer patients who are eligible for endocrine therapy with ARTA plus LHRH agonist.
  Interventions: Diagnostic Test: Periodic ARV7 and miRNA evaluation

INTERVENTIONS:
Diagnostic Test: Periodic ARV7 and miRNA evaluation — Determination of AR-V7 splice variants on circulating tumor cells and evaluation of circulating levels of miRNA by blood sample collection during PSA assessment at different time points along the treatment course (initiation, 8-weeks assessment, progression).

SUMMARY:
Observational prospective study investigating the plasmatic levels of miRNA according to AR-V7 mutational status in mCRPC patients receiving standard of care therapy. At the time of the enrollment, patients will undergo determination of AR-V7 splice variants on circulating tumor cells and periodic assessment of circulating levels of miRNA at different time points during the treatment course (initiation, 8-weeks assessment, progression); irrespectively of AR-V7 status patients will be allocated to endocrine therapy with enzalutamide or abiraterone plus LHRH agonist (decapeptyl every 3 months) according to standard of care. Integration of local treatment (in particular radiotherapy) will be allowed on oligoprogressive sites of disease and its impact on overall outcome and miRNA levels will be assessed.

DETAILED DESCRIPTION:
Prostate cancer is the most frequent malignancy in male patients; since androgen receptor signalling is capital for cancer progression, androgen deprivation therapy with Luteineizing Hormone Release Hormone Agonists (a LHRH) is the cornerstone of its clinical management until occurrence of castration resistance, resulting in disease relapse following activation of alternative signalling pathways. In order to overcome castration resistance, new generations molecules targeting androgen receptor emerged in the last decade as an alternative to chemotherapy with taxanes: among them Abiraterone and Enzalutamide, a potent androgen receptor inhibitor that restore sensitivity to aLHRH therapy has recently been approved both in the pre-and postchemotherapy setting in metastatic castration-resistant prostate cancer (mCPRC).

Despite promising results, resistance to androgen inhibitors is a critical issue, resulting in treatment failure (primary resistance or adaptative resistance developed during the treatment course), particularly as a result of androgen receptor (AR) amplification or mutations.

This result in a dramatic need to identify predictors of response to treatment in order to choose the correct treatment sequence; nevertheless, this approach is somehow limitated due to scarce avalibility of tissue samples for biomolecular investigation in frail patients with painful bone metastasis.

Among the causes of treatment failure, AR-V7 splice variant of the androgen receptor has been extensively studied by Antonarakis et al, who reported that AR-V7 splice variant in circulating tumor cell (a cost-effective,non invasive assessment performed on blood samples) affects response both to Enzalutamide and to the cytochrome inhibitor Abiraterone, resulting in 0% of PSA response in patients displaying AR-V7(19-39% according to data from Antonarakis et al).

A recent study from Scher et al highlighted that CTC nuclear expression of AR-V7 protein in men with mCRPC as a treatment-specific biomarker was associated with superior survival on taxane therapy over hormone based therapy, advocating for future prospective clinical trials in this setting.

It is therefore most likely that in the next future determination of ARV7 status might become capital in allocating (in almost one third of cases) patients from endocrine therapy to chemotherapy with taxanes;it is also theoretically possible in this scenario that, in case of progression under chemotherapy, those patients considered irreversibly refractory (and thus "lost") to hormone treatment might become eligible to a more and more wide range of genome-driven biologic agents due to increasing availability of genome sequencing techniques that allow to target individual molecular alterations in a tailored perspective.

These future advances might have dramatic consequences on patient management since endocrine therapy as a backbone treatment is a cost-effective, tolerable and safe therapeutic option that should be mantained as long as possible: it is therefore capital to attentively select patient that, despite the presence of an unfavorable biologic profile, maintain a residual sensitivity to hormonal treatment.

It is moreover unclear whether primary resistance could reverse to a more sensitive state: according to recent reports by the same authors AR-V7 positive might revert back to AR-V7 negative status after chemotherapy.

This observation suggest that resistance to endocrine treatment treatment is not an ubiquitous process involving the whole tumor bulk, but arise in most case from clonal expansion of refractory clones in isolated sites of disease progression. In reason of advances in metabolic imaging, these sites could be targeted by locoregional treatment like stereotactic body radiotherapy, a novel radiotherapy modality that allows for focalized delivery of high radiation doses.

In summary, there is an urge to develop new clinical tools to refine patient stratification according to the possibility to extend the use of hormone-based therapies, limiting the resort to chemotherapy and/or biological agents only to selected patients at high risk of progression.

MicroRNA are small non-coding RNAs implicated in protein expression that can be disregulated in various type of cancers. A critical role in prostate cancer progression has been extensively described for:

miRNA 124, a tumor suppressive miRNA, is known to downregulate in vitro the levels of AR transcript variants, as well as alternative signaling networks such as Enhancer of Zeste homolog 2 (EZH2) and Src tyrosine kinase (Src) miR-125b: androgen-independent growth miR-331-3p, miR let-7c, miR-21: transition to castrate-resistant prostate cancer miR-32: androgen-regulated miRNA that is upregulated in CRPC miR-222 : attenuate androgen-induced growth, promote androgen-independent growth miR-30: suppresses ERG expression miR-221, miR-375, and miR-141: overexpressed in metastatic clinically silent cancer MiRNA from peripheral blood samples presents various benefits compared to other techniques, in particular the possibility to assess dynamic changes all along the treatment course to test efficacy of ongoing therapy and the possibility to simultaneously test panels of molecules to identify "signatures" predicting the response to treatment.

HYPOTHESIS Dynamic modifications of circulating miRNA and their correlation with other hallmarks (like presence of AR splice variants) may drive treatment choice and provide valuable informations about response to systemic treatment.

AIM OF THE STUDY To evaluate, in mCRPC patients, a panel of miRNAs involved in various stages of tumor progression and their correlation with AR-V7 mutational status at different time points during the systemic treatment course ( in particular Enzalutamide plus LHRH agonist or Abiraterone plus LHRH agonist or taxane chemotherapy), and their predictive value in terms of response to treatment

STUDY POPULATION Inclusion criteria Castration Resistant Prostate Cancer defined as

* biochemical or clinical progression under therapy with LHRH agonist and
* castrate plasma testosterone levels (<20 ng/dl or <1.73 nmol/L) Eligible for medical treatment Age >18 Informed consentment Exclusion criteria Medical contraindication/refusal to chemotherapy or endocrine therapy Life expectancy inferior to 1 year Previously diagnosed neoplasm

STUDY DESIGN Observational prospective study investigating the plasmatic levels of miRNA according to AR-V7 mutational status in mCRPC patients receiving standard of care therapy. At the time of the enrollment, patients will undergo determination of AR-V7 splice variants on circulating tumor cells and periodic assessment of circulating levels of miRNA at different time points during the treatment course (initiation, 8-weeks assessment, progression); irrespectively of AR-V7 status patients will be allocated to endocrine therapy with enzalutamide or abiraterone plus LHRH agonist (decapeptyl every 3 months) according to standard of care. Integration of local treatment (in particular radiotherapy) will be allowed on oligoprogressive sites of disease and its impact on overall outcome and miRNA levels will be assessed.

STATISTICAL PLAN

Due to the observational nature of the study, we planned a minimum accrual of 45 patients in order to evaluate:

* PSA response (≥50% decline in PSA level from baseline, maintained for ≥4 weeks)
* Best PSA response (maximal percentage decrease in PSA level from baseline )
* Progression-free survival (increase in PSA level ≥ 25% above the nadir )
* Overall survival
* Toxicity (CTCAE V4.0)
* Qol (EORTC QLQ C-30) In the event of disease progression under treatment, in case of oligoprogressive disease (defined as less than 3 sites of disease experiencing progression at restaging imaging ), according to our Institutional practices prosecution of endocrine treatment plus local treatment with radiotherapy will be considered and definitive treatment interruption will be planned in case of further progression 2 months after SBRT.

We envisage a time of accrual of 18 months.

EXPECTED BENEFIT

MiRNA plasma levels might correlate with other predictors of resistance to current standard of care (in particular AR-V7) and may provide real-time information about response to treatment; in the future it may allow to identify subsets of patients that are eligible for integration of systemic therapy with local modalities of treatment to overcome the emergence of refractory clones and maintain durable sensitivity to endocrine treatment and delay the need for chemotherapy even in patients deemed poor-responders.

ELIGIBILITY:
Inclusion Criteria:

* Castration Resistant Prostate Cancer defined as biochemical or clinical progression under therapy with LHRH agonist and castrate plasma testosterone levels (<20 ng/dl or <1.73 nmol/L)
* Eligible for medical treatment
* Age >18 years
* Informed consentment

Exclusion Criteria:

* Medical contraindication/refusal to chemotherapy or endocrine therapy
* Life expectancy inferior to 1 year
* Previously diagnosed neoplasm

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Metastatic castration-resistant prostate cancer (mCPRC) who are eligible for Androgen Receptor Target Agents (Abiraterone Acetate or Enzalutamide) plus LHRH therapy.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Predictive value of miRNA panel in treatment efficacy | 6 months

SECONDARY OUTCOMES:
Comparison predictive value of miRNA and ARV7 status in treatment efficacy | 6 months
Toxicity (CTCAE v.4.03 scale) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Careggi Radiation Oncology Unit, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Result] Egan A, Dong Y, Zhang H, Qi Y, Balk SP, Sartor O. Castration-resistant prostate cancer: adaptive responses in the androgen axis. Cancer Treat Rev. 2014 Apr;40(3):426-33. doi: 10.1016/j.ctrv.2013.09.011. Epub 2013 Sep 14. PMID 24139549
- [Result] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Result] Dehm SM, Schmidt LJ, Heemers HV, Vessella RL, Tindall DJ. Splicing of a novel androgen receptor exon generates a constitutively active androgen receptor that mediates prostate cancer therapy resistance. Cancer Res. 2008 Jul 1;68(13):5469-77. doi: 10.1158/0008-5472.CAN-08-0594. PMID 18593950
- [Result] Efstathiou E, Titus M, Wen S, Hoang A, Karlou M, Ashe R, Tu SM, Aparicio A, Troncoso P, Mohler J, Logothetis CJ. Molecular characterization of enzalutamide-treated bone metastatic castration-resistant prostate cancer. Eur Urol. 2015 Jan;67(1):53-60. doi: 10.1016/j.eururo.2014.05.005. Epub 2014 May 29. PMID 24882673
- [Result] Antonarakis ES, Lu C, Wang H, Luber B, Nakazawa M, Roeser JC, Chen Y, Mohammad TA, Chen Y, Fedor HL, Lotan TL, Zheng Q, De Marzo AM, Isaacs JT, Isaacs WB, Nadal R, Paller CJ, Denmeade SR, Carducci MA, Eisenberger MA, Luo J. AR-V7 and resistance to enzalutamide and abiraterone in prostate cancer. N Engl J Med. 2014 Sep 11;371(11):1028-38. doi: 10.1056/NEJMoa1315815. Epub 2014 Sep 3. PMID 25184630
- [Result] Scher HI, Lu D, Schreiber NA, Louw J, Graf RP, Vargas HA, Johnson A, Jendrisak A, Bambury R, Danila D, McLaughlin B, Wahl J, Greene SB, Heller G, Marrinucci D, Fleisher M, Dittamore R. Association of AR-V7 on Circulating Tumor Cells as a Treatment-Specific Biomarker With Outcomes and Survival in Castration-Resistant Prostate Cancer. JAMA Oncol. 2016 Nov 1;2(11):1441-1449. doi: 10.1001/jamaoncol.2016.1828. PMID 27262168
- [Result] Seisen T, Roupret M, Gomez F, Malouf GG, Shariat SF, Peyronnet B, Spano JP, Cancel-Tassin G, Cussenot O. A comprehensive review of genomic landscape, biomarkers and treatment sequencing in castration-resistant prostate cancer. Cancer Treat Rev. 2016 Jul;48:25-33. doi: 10.1016/j.ctrv.2016.06.005. Epub 2016 Jun 15. PMID 27327958
- [Result] Antonarakis ES, Lu C, Luber B, Wang H, Chen Y, Nakazawa M, Nadal R, Paller CJ, Denmeade SR, Carducci MA, Eisenberger MA, Luo J. Androgen Receptor Splice Variant 7 and Efficacy of Taxane Chemotherapy in Patients With Metastatic Castration-Resistant Prostate Cancer. JAMA Oncol. 2015 Aug;1(5):582-91. doi: 10.1001/jamaoncol.2015.1341. PMID 26181238
- [Result] Nakazawa M, Lu C, Chen Y, Paller CJ, Carducci MA, Eisenberger MA, Luo J, Antonarakis ES. Serial blood-based analysis of AR-V7 in men with advanced prostate cancer. Ann Oncol. 2015 Sep;26(9):1859-1865. doi: 10.1093/annonc/mdv282. Epub 2015 Jun 27. PMID 26117829
- [Result] Hellman S, Weichselbaum RR. Importance of local control in an era of systemic therapy. Nat Clin Pract Oncol. 2005 Feb;2(2):60-1. doi: 10.1038/ncponc0075. No abstract available. PMID 16264859
- [Result] Shi XB, Ma AH, Xue L, Li M, Nguyen HG, Yang JC, Tepper CG, Gandour-Edwards R, Evans CP, Kung HJ, deVere White RW. miR-124 and Androgen Receptor Signaling Inhibitors Repress Prostate Cancer Growth by Downregulating Androgen Receptor Splice Variants, EZH2, and Src. Cancer Res. 2015 Dec 15;75(24):5309-17. doi: 10.1158/0008-5472.CAN-14-0795. Epub 2015 Nov 16. PMID 26573802
- [Result] Shi XB, Xue L, Ma AH, Tepper CG, Kung HJ, White RW. miR-125b promotes growth of prostate cancer xenograft tumor through targeting pro-apoptotic genes. Prostate. 2011 Apr;71(5):538-49. doi: 10.1002/pros.21270. Epub 2010 Sep 30. PMID 20886540
- [Result] Epis MR, Giles KM, Barker A, Kendrick TS, Leedman PJ. miR-331-3p regulates ERBB-2 expression and androgen receptor signaling in prostate cancer. J Biol Chem. 2009 Sep 11;284(37):24696-704. doi: 10.1074/jbc.M109.030098. Epub 2009 Jul 7. PMID 19584056
- [Result] Yang CH, Yue J, Fan M, Pfeffer LM. IFN induces miR-21 through a signal transducer and activator of transcription 3-dependent pathway as a suppressive negative feedback on IFN-induced apoptosis. Cancer Res. 2010 Oct 15;70(20):8108-16. doi: 10.1158/0008-5472.CAN-10-2579. Epub 2010 Sep 2. PMID 20813833
- [Result] Sun T, Wang Q, Balk S, Brown M, Lee GS, Kantoff P. The role of microRNA-221 and microRNA-222 in androgen-independent prostate cancer cell lines. Cancer Res. 2009 Apr 15;69(8):3356-63. doi: 10.1158/0008-5472.CAN-08-4112. Epub 2009 Apr 7. PMID 19351832
- [Result] Kao CJ, Martiniez A, Shi XB, Yang J, Evans CP, Dobi A, deVere White RW, Kung HJ. miR-30 as a tumor suppressor connects EGF/Src signal to ERG and EMT. Oncogene. 2014 May 8;33(19):2495-503. doi: 10.1038/onc.2013.200. Epub 2013 Jun 3. PMID 23728339
- [Result] Brase JC, Johannes M, Schlomm T, Falth M, Haese A, Steuber T, Beissbarth T, Kuner R, Sultmann H. Circulating miRNAs are correlated with tumor progression in prostate cancer. Int J Cancer. 2011 Feb 1;128(3):608-16. doi: 10.1002/ijc.25376. PMID 20473869
- [Result] Waltering KK, Porkka KP, Jalava SE, Urbanucci A, Kohonen PJ, Latonen LM, Kallioniemi OP, Jenster G, Visakorpi T. Androgen regulation of micro-RNAs in prostate cancer. Prostate. 2011 May;71(6):604-14. doi: 10.1002/pros.21276. Epub 2010 Oct 13. PMID 20945501
- [Result] Shen J, Hruby GW, McKiernan JM, Gurvich I, Lipsky MJ, Benson MC, Santella RM. Dysregulation of circulating microRNAs and prediction of aggressive prostate cancer. Prostate. 2012 Sep 15;72(13):1469-77. doi: 10.1002/pros.22499. Epub 2012 Feb 1. PMID 22298119
- [Derived] Francolini G, Loi M, Salvestrini V, Mangoni M, Detti B, Di Cataldo V, Aquilano M, Pinzani P, Salvianti F, Desideri I, Mariotti M, Garlatti P, Stocchi G, Ciccone LP, Lucidi S, Salvatore G, Sottili M, Meattini I, Livi L. Prospective assessment of AR splice variant and PSMA detection on circulating tumor cells of mCRPC patients: preliminary analysis of patients enrolled in PRIMERA trial (NCT04188275). Clin Exp Metastasis. 2021 Oct;38(5):451-458. doi: 10.1007/s10585-021-10118-7. Epub 2021 Aug 19. PMID 34410545
- [Derived] Francolini G, Loi M, Detti B, Desideri I, Mangoni M, Simontacchi G, Meattini I, Livi L. Integrating stereotactic body radiation therapy (SBRT) and systemic treatments in oligoprogressive prostate cancer: new evidence from the literature. Clin Exp Metastasis. 2021 Apr;38(2):227-230. doi: 10.1007/s10585-021-10072-4. Epub 2021 Jan 20. PMID 33471291